CLINICAL TRIAL: NCT06092060
Title: The Effect of a Multi-strain Probiotic Consisting of: Bifidobacterium Lactis W52, Lactobacillus Brevis W63, Lactobacillus Casei W56, Lactococcus Lactis W19, Lactococcus Lactis W58, Lactobacillus Acidophilus W37, Bifidobacterium Bifidum W23, Bifidobacterium Lactis W51, and Lactobacillus Salivarius W24 on Metformin Tolerance and Efficacy With Microbiota and Stool Metabolome in Insulin-resistant Women - a 12-week Randomized, Placebo-controlled, Double-blind Study
Brief Title: The Effect of a Multistrain Probiotic on Metformin Tolerance and Efficacy With Microbiota and Stool Metabolome in Insulin-resistant Women - a 12-week Randomized, Placebo-controlled, Double-blind Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PoznanUPhyEd Probiotyk
Record Dates: First submitted 2023-04-06; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-07

CONDITIONS: Insulin Resistance
Keywords: Insulin Resistance; Multistrain Probiotic; Gut Microbiota
MeSH Terms: conditions — Insulin Resistance | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the group GS (Experimental): probiotic treatment group, ca. 20 participants
  Interventions: Dietary Supplement: the group GS (probiotic)
- the group GP (Placebo Comparator): placebo group, ca. 20 participants
  Interventions: Dietary Supplement: the group GP (placebo)

INTERVENTIONS:
Dietary Supplement: the group GS (probiotic) — The probiotic-supplemented group will receive 2 capsules of freeze-dried powder of a probiotic mixture containing the following bacterial strains twice a day, 3-month: Bifidobacterium lactis W52, Lactobacillus brevis W63, Lactobacillus casei W56, Lactococcus lactis W19, Lactococcus lactis W58, Lactobacillus acidophilus W37, Bifidobacterium bifidum W23, Bifidobacterium lactis W51, Lactobacillus salivarius W24
  Arms: the group GS
Dietary Supplement: the group GP (placebo) — The placebo group will receive 2 capsules consisting of the probiotic product carrier, which is corn starch and maltodextrin, twice a day, 3-month.
  Arms: the group GP

SUMMARY:
The goal of this study is to evaluate the efficacy of metformin on insulin sensitivity and vascular endothelial function with respect to gut microbiota and metabolome in women with established insulin resistance and its tolerance after 12 weeks of probiotic therapy.

The hypothesis is probiotic therapy in women with established insulin resistance undergoing metformin treatment increases the drug's efficacy to improve insulin sensitivity and intestinal endothelial function, and reduces gastrointestinal side effects.

Study participants will be randomly assigned to 2 groups, taking a probiotic (GS) or a placebo (GP). The randomization scheme will be computer-generated using permuted blocks of block size 4.

ELIGIBILITY:
Inclusion Criteria:

* women 25-45 years old, menstruating, BMI 25-32.9 kg / m2, insulin resistance based on the HOMA-IR index (cut-off point 2.5

Exclusion Criteria:

* type 1 and 2 diabetes,
* poorly controlled arterial hypertension (mean SBP values> 140mmHg and / or mean DBP values> 90mmHg) within the last month and / or the need to modify pharmacological treatment,
* 2nd degree obesity, BMI> 35 kg / m2,
* lipid disorders requiring pharmacological treatment in the last 3 months before the start of observation or during observation,
* positive history of ischemic heart disease, carotid and / or lower limb atherosclerosis,
* features of heart failure on physical examination and / or additional examinations (chest X-ray, echocardiography),
* clinically significant arrhythmias or conduction disturbances,
* chronic kidney disease with creatinine clearance <60mL / min / 1.73m2,
* clinically significant impairment of liver function (transaminase values 3 times the normal range),
* acute or chronic, clinically evident inflammatory process (diseases of connective tissue and joints, inflammatory processes of the respiratory tract, inflammatory processes of the genitourinary system, inflammation of the head and neck),
* acute infection in the last month,
* Cancer,
* alcohol abuse, drug addiction,
* taking medications that may interfere with test results,
* Taking antibiotics, steroids, antifungal and antiparasitic agents 4 weeks before the examination (not applicable to topical antifungal agents).
* taking pre - and / or probiotics in the last 12 weeks before the test
* travel to tropical countries in the last 4 weeks prior to the survey
* other conditions that may pose any risk to the patient during the follow-up.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Qualitative assessment of intestinal microbiota in stool samples | up to 10 months
  gut bacteria species in stool will be assessed using the shallow shotgun sequencing method, NGS (Next Generation Sequencing)
Quantitive change in intestinal microbiota in stool samples | up to 10 months
  determination of quantitative (Colony forming units - CFU) changes in bacteria in the stool - the shallow shotgun sequencing method, NGS (Next Generation Sequencing) molecular analysis will be used to assess the changes
Intestinal metabolome in stool samples | up to 10 months
  metabolomic analysis (endogenous metabolism (catabolism of amino acids, lipids), biotransformation products under the influence of xenobiotics (e.g., caffeine), fatty acid biosynthesis, fatty acid derivatives, glycolysis, gluconeogenesis, biosynthesis of primary bile acids, amino acid metabolism, sphingolipid metabolism, unknown metabolites, non-targeted metabolome, short-chain fatty acids) will be performed on a quadrupole mass spectrometer coupled with a time-of-flight (QToF) analyzer connected to the AB Sciex - TripleTOF® 6600+ high performance liquid chromatograph (UHPLC)
Indicators of insulin sensitivity and carbohydrate metabolism | up to 10 months
  Analysis of biochemical indicators related to insulin resistance such as concentrations of glucose, insulin, insulin-like growth factor (IGF-1), hemoglobin A1C (HgA1C), myoglobin
Evaluation of indicators in stool | up to 10 months
  Determination of intestinal inflammatory index - fecal calprotectin, determination of intestinal permeability index - fecal zonulin and determination of intestinal membrane inflammatory index sIgA in feces (RT-PCR and Western blotting).
Indicators of lipid metabolism | up to 10 months
  Concentrations of total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, oxidatively modified LDL lipoprotein (oxLDL), paraoxonase (PON) activity, proprotein convertase subtilisin/kexin 9 (PCSK-9)
Transcription factors regulating carbohydrate and lipid metabolism | up to 10 months
  Peroxisome proliferator-activated receptor (PPARγ; NR1C3), PPARγ coactivator, coactivator 1 α ( PGC -1α)
Adipokines and myokines | up to 10 months
  Analysis of biochemical indicators related to insulin resistance such as leptin, adiponectin, resistin, wisfatin, retinol-binding protein type 4 (RBP4), lipocalin-2, proprotein convertase subtilisin/kexin type 9 (PCSK9)
Indicators of inflammation | up to 10 months
  C-reactive protein (hsCRP), interleukin-1 (IL-1), interleukin-6 (IL-6), interleukin-10 (IL-10), tumor necrosis factor (TNF-alpha), lipocalin-2
Indicators of vascular endothelial function | up to 10 months
  Analysis of biochemical indicators related to insulin resistance and endothelial function, such as endothelial nitric oxide synthase (eNOS), vascular endothelial growth factor (VEGF), homocysteine, plasminogen activator inhibitor 1 (PAI-1), adhesion molecules (sVCAM-1, ICAM-1), monocyte chemoattractant 1(MCP-1), matrix metalloproteinases (MMP-9 and MMP-2), cytosolic fatty acid binding proteins (FABPs)
Indicators of a disrupted intestinal barrier in the blood | up to 10 months
  zonulin, intestinal fatty acid binding protein (I-FABP)

SECONDARY OUTCOMES:
Gastrointestinal disorders questionnaire | up to 10 months
  assessment of gastrointestinal disorders using the Rome IV Questionnaire for adults (selected questions on irritable bowel syndrome, constipation and diarrhea); the statements of the questionnaire relate to frequency and intensity of disorders; higher scores mean worse outcome
Body mass analysis (BMI, kg/m^2) | up to 10 months
  determination of body weight and composition using the electrical bioimpedance method
Body composition analysis (percent of total body mass | up to 10 months
  assessment of bone, fat and fat-free mass using the electrical bioimpedance method
Composite measure of Diet composition assessed by food diaries | up to 10 months
  assessment of protein, fat, carbohydrates, fibre, minerals and vitamins intake using food diaries (grams)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Karolkiewicz, Prof, Principal Investigator — Poznan University of Physical Education
Locations (1):
- Poznan University of Physical Education, Poznan, Poland